CLINICAL TRIAL: NCT07069426
Title: The Effects of Varying Protein Intakes on Muscle Protein Synthesis During Injury-Mediated Muscle Disuse
Brief Title: Muscle Response to Different Amounts of Dietary Protein During Leg Immobilization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 25-04H; MO240092 (Other Grant/Funding Number: MOMRP)
Record Dates: First submitted 2025-05-21; First posted 2025-07-16 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Muscle Disuse; Muscle Disuse Atrophy
Keywords: muscle protein synthesis; muscle disuse; muscle disuse atrophy; immobilization; anabolic resistance; dose-response
MeSH Terms: conditions — Muscular Disorders, Atrophic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Protein Dose (Active Comparator): Participants will consume 20 g of whey protein after 5 days of muscle disuse
  Interventions: Dietary Supplement: 20 grams protein
- High Protein Dose (Active Comparator): Participants will consume 40 g of whey protein after 5 days of muscle disuse
  Interventions: Dietary Supplement: 40 grams protein

INTERVENTIONS:
Dietary Supplement: 20 grams protein — 20 grams of whey protein provided as beverage
  Arms: Standard Protein Dose
Dietary Supplement: 40 grams protein — 40 grams of whey protein provided as beverage
  Arms: High Protein Dose

SUMMARY:
Individuals who sustain musculoskeletal injuries (MSKI) can experience a rapid loss of muscle mass due to declines in muscle loading and activation that occur post-injury (i.e., disuse atrophy). Loss of muscle under these conditions is attributed to a persistent negative net muscle protein balance (muscle protein synthesis [MPS] < muscle protein breakdown) that results, in part, from declines in postprandial MPS (i.e., anabolic resistance). Nutritional interventions that enhance postprandial MPS may be used to overcome disuse-induced anabolic resistance and preserve muscle mass to accelerate recovery and improve recovery outcomes. While supplemental protein has been explored as a potential countermeasure to disuse-induce anabolic resistance, the observed efficacy of such interventions has been mixed. Equivocal findings across studies may be attributed, in part, to an insufficient understanding of what constitutes an effective protein-based intervention. Importantly, no study to date has determined an optimal protein dose for overcoming disuse-induce anabolic resistance, or if there is a threshold for maximally stimulating postprandial MPS under disuse conditions. Therefore, the objective of this work is to determine rates of MPS at rest and in response to standard (20 g) or high (40 g) doses of whey protein during knee immobilization (DISUSE) compared with standard activity (ACTIVE)

DETAILED DESCRIPTION:
Healthy, recreationally active men and women will complete this randomized, double-blind, parallel study. Muscle disuse will be implemented for five days using a unilateral leg immobilization model with one leg assigned to immobilization (DISUSE) and the contralateral leg used as a control (ACTIVE). Immobilization will be implemented with a rigid knee brace fixed at ~60° of flexion and participants will ambulate using crutches. Diets will be standardized during the immobilization phase. Participants will complete a protein feeding study at the end of immobilization consisting of primed, continuous stable isotope infusions, serial blood draws, and muscle biopsies. MPS will be assessed in both the DISUSE and ACTIVE legs in response to standard (20 g) or high (40 g) doses of whey protein. Findings from this work will directly inform the development of targeted nutritional countermeasures for overcoming disuse-induced anabolic resistance and preserving muscle mass after MSKI to optimize physical performance recovery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-39 years (17-39 years if military personnel)
* Body mass index (BMI) between 18.5-32 kg/m2
* Routinely participate in aerobic and/or resistance exercise at least 2 days per week.
* Willing to refrain from alcohol, smoking, smokeless nicotine products (includes e-cigarettes, vaping, chewing tobacco), and dietary supplements (i.e., vitamin D, probiotics) 24 hours before and during immobilization and final testing day.
* Willing to only consume caffeine products provided by study staff during the study.
* Supervisor approval for federal civilian employees and non-SRV active-duty military personnel stationed at NSSC.
* Biological females must have normal menstrual cycles between 26-32 days in duration; 5 menstrual cycles within the past 6 months; or on continuous hormonal contraception (i.e., IUD or oral contraceptives without placebo).

Exclusion Criteria:

* Musculoskeletal injuries that may interfere with the safe use of crutches.
* Personal or family history of thrombosis, or prior diagnosis of deep vein thrombosis (DVT) or pulmonary embolism (PE).
* Metabolic or cardiovascular abnormalities, gastrointestinal disorders, neuromuscular disorders, lower-limb amputation, or muscle/bone wasting disorders (e.g., diabetes, cardiovascular disease, Crohn's disease, etc.).
* Taking medication that affects macronutrient utilization (i.e., statins, corticosteroids, weight loss medications such as Ozempic, etc.).
* Significantly abnormal blood clotting as determined by USARIEM Office of Medical Oversight (OMSO) or home duty station medical support (HMS).
* Allergy to lidocaine (or similar local anesthetic).
* Present condition of alcoholism, anabolic steroid use, or other substance abuse issues as determined by OMSO or HMS.
* Blood donation within 8-wk of beginning the study.
* Pregnant, trying to become pregnant, and/or breastfeeding (results of urine pregnancy test and self-report for breastfeeding will be obtained before body composition testing).
* Unwilling or unable to consume study diets or foods provided due to personal preference and/or food allergies.
* Unwilling or unable to adhere to study physical restrictions (i.e., no structured physical activity or recreational activity beyond activities of daily living) 24 hours before and during immobilization, and the final testing day.
* Unwilling or unable to keep the knee brace on and walk with crutches during the immobilization phase.

Ages: 17 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Rates of postabsorptive and postprandial muscle protein synthesis assessed using 2H5-Phenylalanine stable isotope methodologies. | After 5 days of muscle disuse
  Postabsorptive and postprandial muscle protein synthesis in response to 20 or 40 g of whey protein determined using 2H5-Phenylalanine stable isotope methodologies and expressed as fractional synthetic rate (FSR).

CONTACTS AND LOCATIONS:
Locations (1):
- US Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.